CLINICAL TRIAL: NCT06121583
Title: Cross-sectional, Non-randomized Observational Study to Assess the Frequency of Reduced Sodium Intake in the Primary Care Setting - LAXAP
Acronym: LAXAP
Status: Completed | Type: Observational
Sponsor: Casen Recordati S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAXAP-CASEN-NI 0600
Record Dates: First submitted 2023-10-31; First posted 2023-11-08 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Dietary Deficiency; Sodium
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a cross-sectional epidemiological, observational study. It would be carried out in primary health care sites. The purpose of this study is estimating the percentage of patients aged 60 years or older who suffer from a condition, or take medication, associated with a low or sodium-free diet in primary care consultations.

This is a cross-sectional epidemiological study of data collection without medication.

Participants data will be collected after obtaining their confirmation through an Informed Consent From. No medication will be given to patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the primary care unit, in person, with inclusion beginning in order of care in consultation from the beginning of the study.
* Age greater than or equal to 60 years.

Exclusion Criteria: Not applicable

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (over 60 years of age or older) who attend primary care units
Sampling Method: Non-Probability Sample
Enrollment: 449 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who suffer from a condition or take medication associated with a diet low or absent of sodium. | At the time of the consultation, anticipated average 1 hour
  Patients who require to follow a diet with low sodium content defined as patients that suffer from a condition or take medication associated with a diet low or absent of sodium:
  Right or congestive heart failure, Acute kidney failure, Chronic renal failure, Nephrotic syndrome, Edematogenic glomerulonephritis, Diabetic nephropathy, Nephrolithiasis, Arterial hypertension, Ascites, Hepatic cirrhosis, Prolonged treatments (more than 6 months) with corticosteroids

SECONDARY OUTCOMES:
Percentage of patients who present a recommendation/prescription for a low-sodium diet. | At the time of the consultation, anticipated average 1 hour
Percentage of patients with constipation | At the time of the consultation, anticipated average 1 hour
  Constipation according to Rome III: a diagnosis of functional constipation is made when at least two of the following criteria are met for the last 3 months with symptom onset at least 6 months prior to diagnosis: a) straining on >25% of defecations; b) lumpy or hard stools on >25% of defecations; c) sensation of incomplete evacuation on >25% of defecations; d) sensation of anorectal obstruction/blockage on >25% of defecations; e) manual maneuvers on >25% of defecations; and f) less than 3 defecations per week.
Percentage of patients who take laxatives | At the time of the consultation, anticipated average 1 hour
Percentage of patients who present constipation and suffer from a condition or take medication associated with a diet low or absent of sodium. | At the time of the consultation, anticipated average 1 hour
  Constipation according to Rome III: a diagnosis of functional constipation is made when at least two of the following criteria are met for the last 3 months with symptom onset at least 6 months prior to diagnosis: a) straining on >25% of defecations; b) lumpy or hard stools on >25% of defecations; c) sensation of incomplete evacuation on >25% of defecations; d) sensation of anorectal obstruction/blockage on >25% of defecations; e) manual maneuvers on >25% of defecations; and f) less than 3 defecations per week.
  Patients who require to follow a diet with low sodium content defined as patients that suffer from a condition or take medication associated with a diet low or absent of sodium:
  Right or congestive heart failure, Acute kidney failure, Chronic renal failure, Nephrotic syndrome, Edematogenic glomerulonephritis, Diabetic nephropathy, Nephrolithiasis, Arterial hypertension, Ascites, Hepatic cirrhosis, Prolonged treatments (more than 6 months) with corticosteroids
Percentage of patients who present constipation and suffer from a condition or take a medication associated with a low or absent sodium diet and receive a prescription for a laxative with a high level of sodium | At the time of the consultation, anticipated average 1 hour
  Constipation according to Rome III: a diagnosis of functional constipation is made when at least two of the following criteria are met for the last 3 months with symptom onset at least 6 months prior to diagnosis: a) straining on >25% of defecations; b) lumpy or hard stools on >25% of defecations; c) sensation of incomplete evacuation on >25% of defecations; d) sensation of anorectal obstruction/blockage on >25% of defecations; e) manual maneuvers on >25% of defecations; and f) less than 3 defecations per week.
  Patients who require to follow a diet with low sodium content defined as patients that suffer from a condition or take medication associated with a diet low or absent of sodium:
  Right or congestive heart failure, Acute kidney failure, Chronic renal failure, Nephrotic syndrome, Edematogenic glomerulonephritis, Diabetic nephropathy, Nephrolithiasis, Arterial hypertension, Ascites, Hepatic cirrhosis, Prolonged treatments (more than 6 months) with corticosteroids
Percentage of patients with each of the diseases or taking treatments that recommend the intake of a diet with low sodium content. | At the time of the consultation, anticipated average 1 hour
  Patients that suffer from a condition or take medication associated with a diet low or absent of sodium:
  Right or congestive heart failure, Acute kidney failure, Chronic renal failure, Nephrotic syndrome, Edematogenic glomerulonephritis, Diabetic nephropathy, Nephrolithiasis, Arterial hypertension, Ascites, Hepatic cirrhosis, Prolonged treatments (more than 6 months) with corticosteroids
Percentage of patients who have sodium restriction in the diet and receive sodium in the form of concomitant medication. | At the time of the consultation, anticipated average 1 hour
Description of each of the study populations | At the time of the consultation, anticipated average 1 hour
  Description of patients who suffer from a condition or take a medication associated with a low or no sodium diet, patients with a low sodium diet recommendation, patients with constipation, patients taking laxatives: Data demographics, anthropometric data, diseases associated with a low sodium diet, constipation, laxatives and concomitant medication. In terms of their demographics and clinical characteristics.
Percentage of patients with concomitant medication that may affect the amount of sodium in the blood by type, dosage, duration of treatment | At the time of the consultation, anticipated average 1 hour

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Centro de Salud Just Oliveras, L'Hospitalet de Llobregat, Barcelona
  - Centro de Salud Gracia Sabadell, Sabadell, Barcelona
  - Centro de Salud La Barrera, Castro Urdiales, Cantabria
  - Consultorio Ojo de Garza, Las Palmas de Gran Canaria, Gran Canaria
  - Centro de Salud Reyes Magos, Alcalá de Henares, Madrid
  - Centro de Salud Abarán, Abarán, Murcia
  - Centro de Salud Cieza Este, Cieza, Murcia
  - Centro de Salud Dr. Guigou, Santa Cruz de Tenerife, Tenerife
  - Centro de Salud Icod de los Vinos, Santa Cruz de Tenerife, Tenerife
  - Centro de Salud Adrià, Barcelona
  - Centro de Salud Avenida de Aragón, Madrid
  - Centro de Salud Daroca, Madrid
  - Centro de Salud Goya, Madrid
  - Centro de Salud Potes, Madrid

IPD SHARING:
Plan to Share IPD: No
there is no IMPD object of the study